CLINICAL TRIAL: NCT03071588
Title: Assessment of a New Protocol for Indirect Pulp Capping Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14/LO/0880
Record Dates: First submitted 2017-02-23; First posted 2017-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Reversible Pulpitis

STUDY DESIGN:
Intervention Model Description: Two groups of patients, each group received the investigated intervention at baseline and being followed up in parallel for one year.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): the conventional protocol in indirect pulp capping include the use of mechanical rotary burs for caries removal in teeth with reversible pulpitis.
  Interventions: Device: Mechanical rotary burs
- Conservative (Experimental): the conservative protocol of indirect pulp capping include the use of Carisolv gel for caries removal in teeth with reversible pulpitis.
  Interventions: Device: Carisolv gel

INTERVENTIONS:
Device: Mechanical rotary burs — A rotary drill made of steel or diamond impregnated materials attached to a steel shank, available in varying degree of sharpness, lengths and sizes used conventionally in preparation of teeth to receive a dental restoration.
  Arms: Control
Device: Carisolv gel — A chemical gel made of a combination of amino acids and sodium hypochlorite used with hand instruments to soften and remove the decay to prepare the tooth to receive a dental restoration.
  Arms: Conservative

SUMMARY:
The aim of the study is to assess clinically, radiographically and microbiologically a new protocol for indirect pulp capping procedures compared to the conventional protocol in painful teeth. It was postulated that there is no difference between both protocols in terms clinical, radiographical and microbial outcome measure after one year of follow up in painful teeth.

DETAILED DESCRIPTION:
Indirect pulp capping is a common dental procedure carried out on painful teeth with deep cavities resulting from dental decay in an attempt to prolong the life of the tooth / pulp while relieving pain, This study aims primarily to assess the response of the pulp of the tooth to two different clinical procedures used in the treatment of deep caries. One group of patients will be treated with a standard clinical procedure which involve mechanical rotary burs with no magnification for caries removal, the other group will be treated with a more conservative clinical procedure using CarisolvTM gel with the aid of an operating microscope for caries removal. The study also involves taking of samples from the tooth decay for microbiological / biochemical analysis and evaluation to determine the species richness in the bacterial community associated with this condition. The study also compare the radiographical findings of 3D cone beam computed tomography (CBCT) scans with that of normal Xrays in detecting the presence of early bone changes associated with the roots of these teeth.

The study carried out at King's College London/ Dental Institute at Guy's Hospital and form part of the routine dental treatment done at the emergency dental clinics with the exception of the CBCT scans. Volunteers given written information about the process and given time to consider participation. Once any questions have been answered, fully informed written consent obtained if they are interested in taking part. At least one deep cavity causing toothache requiring indirect pulp capping detected and diagnosed through conventional clinical and Xray dental assessment. The procedure involves removal of the decay using one of the proposed clinical techniques and the placement of a pulp capping material according to manufacturer's instructions and the definitive filling will be placed, follow up will at 12 months. Radiographic assessment including cone beam computed tomography (CBCT) will be done at baseline and 12 months. It is hoped that data analysed from this study will provide a definitive clinical and radiographic evidence base for the outcome of the indirect pulp capping operative treatment procedure.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of reversible pulpitis with positive response to cold pulp test.

Exclusion Criteria:

Clinical diagnosis of irreversible pulpitis, Pregnant women, mobile teeth and teeth with tenderness to percussion.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
cold pulp test (signalling the nerve of the pulp of the tooth by cold application) | One year follow up
  Binary variable outcome measure whether the nerve is positively or negatively responsive to the cold test.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Mannocci, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali AH, Thani FB, Foschi F, Banerjee A, Mannocci F. Self-Limiting versus Rotary Subjective Carious Tissue Removal: A Randomized Controlled Clinical Trial-2-Year Results. J Clin Med. 2020 Aug 25;9(9):2738. doi: 10.3390/jcm9092738. PMID 32854206
- [Derived] Ali AH, Koller G, Foschi F, Andiappan M, Bruce KD, Banerjee A, Mannocci F. Self-Limiting versus Conventional Caries Removal: A Randomized Clinical Trial. J Dent Res. 2018 Oct;97(11):1207-1213. doi: 10.1177/0022034518769255. Epub 2018 May 8. PMID 29738286